CLINICAL TRIAL: NCT03522922
Title: Efficacy of Microneedling With Topical Vitamin C in Treatment of Acne Scarring
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rasha Ismail, Assistant lecturer, Department of Dermatology, Venereology and Andrology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNC.001
Record Dates: First submitted 2018-03-04; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Acne Vulgaris; Acne Scars
Keywords: Acne scars; dermaroller; vitamin C
MeSH Terms: conditions — Acne Vulgaris | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dermaroller arm (Active Comparator): Patients received a series of six treatments by dermaroller at 4 weeks interval and no topical anti scar treatment in between sessions.
  Interventions: Device: Dermaroller
- Dermaroller + topical Vit. C arm (Active Comparator): Patients received a series of six treatments by dermaroller at 4 weeks interval with the same maneuver and instructions as first group and each session was followed by immediate application of topical vitamin C serum plus once daily application in between sessions.
  Interventions: Device: Dermaroller; Drug: Topical Vitamin C
- Topical Vit. C arm (Active Comparator): Patients received once daily topical vitamin C serum capsule at night for six months. With monthly evaluation.
  Interventions: Drug: Topical Vitamin C

INTERVENTIONS:
Device: Dermaroller — The derma roller used (dermaroller MF8, MT dermaroller Beverly Hills, California USA) is a plastic device with a 12-cm handle that holds a drum-shaped cylinder at the end, similar to a small paint roller, 2 cm in diameter and 2 cm in width. The surface of the cylinder holds 192 titanium needles in eight rows. Each 0.25 mm in diameter and 1.5 mm length sterilized by UV/ Gamma rays.
  Arms: Dermaroller + topical Vit. C arm; Dermaroller arm
Drug: Topical Vitamin C — The used vitamin C product was in the form of 17% concentration of L- Ascorbic Acid serum that was encapsulated in gelatinous capsules each contain 1 mg of the serum. The patient instructed to open one capsule and apply its serum content on the treatment area daily at night. This capsule form for topical application help to insure stability of the product and also insure use of equal dose in each application
  Other Names: Topical Vit.C
  Arms: Dermaroller + topical Vit. C arm; Topical Vit. C arm

SUMMARY:
This study aimed to evaluate the efficacy of dermaroller and topical vitamin C- either separate or combined- in treatment of post acne scars.

prospective randomized clinical trial that was The study was a randomized controlled trial, conducted in Sohag Dermatology outpatient clinic between June 2016 and of February 2018. 30 patients with acne scars were included.

All patients were informed about the entire procedure, medication, possible side effects and outcomes. A written informed consent was signed from each participant.

DETAILED DESCRIPTION:
Study population:

Each study group included 10 patients. Detailed history and full clinical examination was conducted for each patient. Patients had 6 visits at one month interval to receive treatment and evaluated one month after the end of treatment visits.

The first group:

Patients received a series of six treatments by dermaroller at 4 weeks interval and no topical anti scar treatment in between sessions.

The second group:

Received a series of six treatments by dermaroller at 4 weeks interval with the same maneuver and instructions as first group and each session was followed by immediate application of topical vit.C serum plus once daily application in between sessions.

The third group:

received once daily topical vit.C serum capsule at night for six months. With monthly evaluation.

Assessment of patients during visits was as follow:

A) Clinical evaluation by B) Photographic documentation C) Patient satisfaction D) Safety assessment

ELIGIBILITY:
Inclusion Criteria:

* Facial acne scars

Exclusion Criteria:

* Active inflammatory acne.
* Active infection in the treatment area (e.g., herpes simplex and verrucae).
* Melanoma or lesions suspected of malignancy.
* Isotretinoin use in the past year.
* Dermatoses (e.g., eczema and psoriasis).
* Sunburn.
* Anticoagulant therapy.
* Systemic disease (diabetes, hypertension, collagen disease or bleeding tendency).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical response by (ECCA) scale | 9 months
  Assessment of clinical response before intervention,after each session and at monthly intervals for 3 months after the end of sessions. Echellad'e valuation Clinique des cicatrices d'acne (ECCA) scale was used for numerical grading of acne scars.The ECCA grading scale is a tool designed to help dermatologists to assess the severity of acne scars and to standardize the discussions about the treatments of scars. The scale grades from no scar (grade = 0) to many scars (grade= 3)

SECONDARY OUTCOMES:
Patient satisfaction questionnaire | 9 months
  Patient satisfaction at the end of study graded as one of four categories represents the % of subjective improvement in the acne scars after treatment as compared with prior to treatment: [(Excellent (100% -76%)- Very Good (51% - 75%) -good (26% - 50%)- poor (0% - 25%)]

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan Saleh, MD, Study Director — Sohag Faculty of Medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Share any information about the study with other researchers after acceptance of all authors.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available by the end of April 2018, without time frame.
Access Criteria: To all interested researchers